CLINICAL TRIAL: NCT00401830
Title: A Parallel, Randomized, Double-Blind, Placebo-Controlled, Multicenter Proof of Concept Trial to Assess the Efficacy and Safety of 400 mg/Day Lacosamide Tablets in Subjects With Signs and Symptoms Associated With Fibromyalgia Syndrome
Brief Title: Assessing Efficacy and Safety of Lacosamide Compared to Placebo in Reducing Signs and Symptoms of Fibromyalgia Syndrome.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP0887
Expanded Access: NCT03559673 (No longer available)
Record Dates: First submitted 2006-11-09; First posted 2006-11-22 (Estimated); Results first posted 2009-10-22 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2017-07

CONDITIONS: Fibromyalgia Syndrome
Keywords: Fibromyalgia Syndrome; Lacosamide; Vimpat; Harkoseride
MeSH Terms: conditions — Fibromyalgia | interventions — Lacosamide; 2-(acetylamino)-3-methoxy-N-(phenylmethyl)-, (2R)-

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Lacosamide (Experimental): Lacosamide Tablet 400mg daily
  Interventions: Drug: Lacosamide

INTERVENTIONS:
Drug: Lacosamide — Tablet 400mg daily (200mg twice daily) during 8-week maintenance phase following 4-week titration phase starting at 100mg/day and increasing to 400mg/day at weekly intervals of 100mg
  Other Names: Vimpat; Harkoseride
  Arms: Lacosamide
Other: Placebo — Matching placebo tablet administered twice daily
  Arms: Placebo

SUMMARY:
This trial investigated the efficacy and safety of 400mg/day of lacosamide as compared to placebo in reducing the signs and symptoms of fibromyalgia syndrome.

DETAILED DESCRIPTION:
This was a proof-of-concept study and not powered for statistical comparisons.

The trial consisted of a 4-week Titration Phase, an 8-week Maintenance Phase, a 1-week Taper Phase, and a 2-week Safety Follow-Up Phase. If subjects met the eligibility criteria, they were randomized to receive either lacosamide 400mg/day or placebo during the Maintenance Phase. Subjects assigned to lacosamide were titrated from 100mg/day to 400mg/day at weekly intervals of 100mg. All subjects who completed the 4-week Titration Phase entered an 8-week Maintenance Phase. No dose adjustment was allowed during the Maintenance Phase. The Treatment Phase was defined as the combined Titration and Maintenance Phases.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, 18 to 65 years old
* Fulfills all 3 points of American College of Rheumatology (ACR) definition for diagnosis of fibromyalgia
* At least moderate pain (pain intensity ≥ 5 on Likert pain scale (0-10) during the 7 days prior to Baseline)
* Fibromyalgia Impact Questionnaire (FIQ) total score ≥ 50
* Completed an adequate washout period for excluded medications prior to beginning the Baseline Diary Phase

Exclusion Criteria:

* Symptomatic regional or structural rheumatic disease
* Diagnosed neuropathic pain syndrome
* Receiving treatment with neurostimulating devices
* Significant psychopathology
* History of chronic alcohol or drug abuse within 6 months prior to Screening
* Been hospitalized for psychiatric or behavioral reasons within 6 months prior to Screening
* Clinically significant abnormal vitals, cardiac dysfunction and /or arrhythmias
* Taken neuroleptics, serotonin and norepinephrine reuptake inhibitors (SNRIs) or tricyclic antidepressants (TCAs)
* Other medical conditions that could compromise the subject's ability to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2006-10; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (24):
- United States (24):
  - Litchfield Park, Arizona
  - Santa Ana, California
  - Walnut Creek, California
  - Deerfield Beach, Florida
  - Fort Lauderdale, Florida
  - Fort Myers, Florida
  - Tampa, Florida
  - Athens, Georgia
  - Decatur, Georgia
  - Peoria, Illinois
  - Evansville, Indiana
  - Madisonville, Kentucky
  - Columbia, Maryland
  - Frederick, Maryland
  - Brockton, Massachusetts
  - Charlotte, North Carolina
  - Winston-Salem, North Carolina
  - Mogadore, Ohio
  - Toledo, Ohio
  - Goose Creek, South Carolina
  - Memphis, Tennessee
  - San Antonio, Texas
  - Richmond, Virginia
  - Kirkland, Washington

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Matching placebo tablet (administered twice daily)
- Lacosamide: Lacosamide Tablet 400mg daily (administered twice daily)
Period: Overall Study
Arm/Group | Placebo | Lacosamide
Started | 81 | 78
Completed | 50 | 46
Not Completed | 31 | 32
Not completed — Adverse Event | 10 | 18
Not completed — Lack of Efficacy | 11 | 5
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Protocol Violation | 3 | 3
Not completed — Non-compliance with drug study | 1 | 0
Not completed — Lost to Follow-up | 1 | 3
Not completed — Other: Personal / Family problems | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Lacosamide | Total
Number analyzed (Participants) | 81 | 78 | 159
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 79 | 76 | 155
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (10.5) | 48.9 (11.1) | 49.7 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 71 | 148
  Male | 4 | 7 | 11
Region of Enrollment [Number; unit: participants]
  United States | 81 | 78 | 159

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Daily Pain Score to the Last 2 Weeks of the 12-week Treatment Phase (Based on the Full Analysis Set)
Description: The average daily pain score is calculated using an 11-point Likert scale, ranging from 0 (no pain) to 10 (worst pain ever experienced).
Time Frame: Baseline, Last 2 weeks of the 12-week Treatment Phase
Population: Of the 81 (Placebo) and 78 (Lacosamide) patients randomized, 80 and 78 patients respectively are included in the summary of the last 2 weeks of the 12-week Treatment Phase, based on the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Lacosamide
Number analyzed (Participants) | 80 | 78
Score on a scale | -1.30 (1.92) | -1.80 (2.13)

2. Primary Outcome: Change From Baseline in Average Daily Pain Score to the Last 2 Weeks of the 12-week Treatment Phase (Based on the Per Protocol Set)
Description: as for outcome 1
Time Frame: Baseline, Last 2 weeks of the 12-week Treatment Phase
Population: Of the 81 (Placebo) and 78 (Lacosamide) patients randomized, 36 and 41 patients respectively are included in the summary of the last 2 weeks of the 12-week Treatment Phase, based on the Per Protocol Set.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Lacosamide
Number analyzed (Participants) | 36 | 41
Score on a scale | -2.11 (1.98) | -2.40 (2.08)

3. Secondary Outcome: Change From Baseline in Fibromyalgia Impact Questionnaire (FIQ) Total Score to the Last Assessment in the 12-week Treatment Phase
Description: The Fibromyalgia Impact Questionnaire (FIQ) Total Score ranges from 0 to 100 with higher scores corresponding to a greater impact of fibromyalgia
Time Frame: Baseline, Last assessment in the 12-week Treatment Phase
Population: Of the 81 (Placebo) and 78 (Lacosamide) patients randomized, 79 and 78 patients respectively are included in this summary based on the Full Analysis Set and have the Last Assessment in the 12-week Treatment Phase.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Lacosamide
Number analyzed (Participants) | 79 | 78
Score on a scale | -14.7 (16.9) | -17.5 (19.3)

4. Secondary Outcome: Change From Baseline in Total Myalgic Score to the Last Assessment in the 12-week Treatment Phase
Description: Total Myalgic Score ranges from 0 to 54 with higher scores corresponding to a greater level of pain.
Time Frame: Baseline, Last assessment in the 12-week Treatment Phase
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Lacosamide
Number analyzed (Participants) | 79 | 78
Score on a scale | -6.7 (13.6) | -9.7 (13.0)

5. Secondary Outcome: Change From Baseline in Average Daily Interference With Sleep to the Last 2 Weeks of the 12-week Treatment Phase
Description: Sleep scale - the subject rated quality of sleep, from 0 (very good sleep) to 10 (very poor sleep)
Time Frame: Baseline, Last 2 weeks of the 12-week Treatment Phase
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Lacosamide
Number analyzed (Participants) | 80 | 78
Score on a scale | -1.24 (1.94) | -1.64 (2.16)

6. Secondary Outcome: Change From Baseline in Daily Interference With General Activity to the Last 2 Weeks of the 12-week Treatment Phase
Description: General activity scale - the subject rated how the pain had interfered with general activity, from 0 (did not interfere) to 10 (completely interfered)
Time Frame: Baseline, Last 2 weeks of the 12-week Treatment Phase
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Lacosamide
Number analyzed (Participants) | 80 | 78
Score on a scale | -1.27 (1.93) | -1.44 (2.30)

7. Secondary Outcome: Change From Baseline in Morning Pain Score to the Last 2 Weeks of the 12-week Treatment Phase
Description: An 11-point Likert scale was used for subjects to assess pain, from 0 (no pain) to 10 (worst pain ever experienced).
Time Frame: Baseline, Last 2 weeks of the 12 week Treatment Phase
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Lacosamide
Number analyzed (Participants) | 80 | 78
Score on a scale | -1.29 (1.97) | -1.77 (2.18)

8. Secondary Outcome: Change From Baseline in Evening Pain Score to the Last 2 Weeks of the 12-week Treatment Phase
Description: An 11-point Likert scale was used for subjects to assess pain, from 0 (no pain) to 10 (worst pain ever experienced).
Time Frame: Baseline, Last 2 weeks of the 12 week Treatment Phase
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Lacosamide
Number analyzed (Participants) | 80 | 78
Score on a scale | -1.32 (1.94) | -1.84 (2.15)

9. Secondary Outcome: Patient Global Impression of Change (PGIC) Assessment From Baseline to the Last Assessment in the 12-week Treatment Phase
Description: The PGIC is a 7-point self-administered categorical rating scale in which the subject rated the change in pain since starting trial medication (from much worse [score of 1] to much better [score of 7]).
Time Frame: Baseline, Last assessment in the 12-week Treatment Phase
Population: Of the 81 (Placebo) and 78 (Lacosamide) patients randomized, 80 and 78 patients respectively are included in the Full Analysis Set (FAS). A total of 67 subjects in each treatment group in the FAS have this assessment.
Measure: Number; unit: Patients
Arm/Group | Placebo | Lacosamide
Number analyzed (Participants) | 67 | 67
Patients
  Much better | 8 | 17
  Moderately better | 14 | 12
  Mildly better | 18 | 13
  No change | 17 | 13
  Mildly worse | 5 | 3
  Moderately worse | 2 | 6
  Much worse | 3 | 3

10. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HADS) Scores to the Last Assessment in the 12-week Treatment Phase
Description: The Hospital Anxiety and Depression Scale (HADS) is a self-administered instrument for detecting anxiety and depression in medical outpatients. Scores range from 0 to 21 for each subscale with higher scores reflecting a greater level of anxiety or depression.
Time Frame: Baseline, Last assessment in the 12-week Treatment Phase
Population: Of the 81 (Placebo) and 78 (Lacosamide) patients randomized, 80 and 78 patients respectively are included in the Full Analysis Set (FAS). A total of 67 subjects in each treatment group in the FAS have change from Baseline data for depression. One subject in the Lacosamide group had a missing anxiety score.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Lacosamide
Number analyzed (Participants) | 67 | 67
Score on a scale
  Depression score (Placebo n=67, Lacosamide n=67) | -1.1 (2.8) | -0.8 (2.8)
  Anxiety Score (Placebo n=67, Lacosamide n=66) | -1.2 (3.2) | -1.2 (3.2)

11. Secondary Outcome: Percentage of Patients Using Rescue Medication During the 12-week Treatment Phase
Description: Subjects recorded use of rescue medication for pain in the diary daily in the evening with a Yes/No response.
Time Frame: 12-week Treatment Phase
Population: Of the 81 (Placebo) and 78 (Lacosamide) patients randomized, 80 and 78 patients respectively are included in this summary based on the Full Analysis Set.
Measure: Number; unit: Percentage of patients
Arm/Group | Placebo | Lacosamide
Number analyzed (Participants) | 80 | 78
Percentage of patients | 83.8 | 83.3

12. Secondary Outcome: Percentage of Patients Using Alcohol for Pain During the 12-week Treatment Phase
Description: Use of alcohol to treat pain in the past 24 hours was recorded (Yes/No response).
Time Frame: 12-week Treatment Phase
Population: as for outcome 11
Measure: Number; unit: Percentage of patients
Arm/Group | Placebo | Lacosamide
Number analyzed (Participants) | 80 | 78
Percentage of patients | 17.5 | 15.4

13. Secondary Outcome: Change From Baseline in Fibromyalgia Symptom Scores to the Last Assessment in the 12-week Treatment Phase
Description: All scores range from 0 to 10 with higher scores corresponding to a greater level of symptom severity.
Time Frame: Baseline, Last assessment in the 12-week Treatment Phase
Population: Of the 81 (Placebo) and 78 (Lacosamide) patients randomized, 61 and 60 patients respectively are included in this summary based on the Full Analysis Set and have the Last Assessment in the 12-week Treatment Phase.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Lacosamide
Number analyzed (Participants) | 61 | 60
Score on a scale
  Muscular Pain | -1.9 (2.4) | -2.4 (2.9)
  Fatigue | -1.7 (2.4) | -1.9 (2.9)
  Insomnia | -1.9 (2.7) | -2.4 (3.2)
  Joint pains | -1.9 (2.8) | -1.9 (3.3)
  Headaches | -0.7 (3.2) | -1.2 (3.5)
  Restless legs | -1.5 (2.9) | -1.2 (3.3)
  Paresthesias | -1.6 (2.6) | -1.3 (3.1)
  Impaired memory | -1.3 (2.7) | 0.0 (3.1)
  Leg cramps | -1.5 (2.8) | -1.4 (2.8)
  Impaired concentration | -1.2 (3.1) | -0.5 (3.1)
  Abdominal pain, alternating diarrhea/constipation | -1.7 (3.4) | -1.2 (3.5)

14. Secondary Outcome: Lacosamide Plasma Concentration at the End of the Maintenance Phase/ Week 12
Time Frame: End of the Maintenance Phase/Week 12
Population: The number of patients in the Placebo treatment group has been presented as 0 as this outcome measure is not applicable for this treatment group. Of the 78 patients in the Lacosamide treatment group (Safety Set) data were available at the end of Maintenance Phase/Week 12 for the 45 patients remaining in the study.
Measure: Mean (Standard Deviation); unit: ug/ML
Arm/Group | Placebo | Lacosamide
Number analyzed (Participants) | 0 | 45
ug/ML |  | 9.44 (5.24)

ADVERSE EVENTS:
Arm/Group | Placebo | Lacosamide
Serious Adverse Events (participants affected / at risk) | 3/81 | 0/78
Other Adverse Events (participants affected / at risk) | 37/81 | 53/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=81) | Lacosamide (N=78)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=81) | Lacosamide (N=78)
Vision blurred (Eye disorders) | 1 (1) | 4 (5)
Constipation (Gastrointestinal disorders) | 3 (3) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 6 (7) | 5 (5)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 4 (4)
Nausea (Gastrointestinal disorders) | 12 (13) | 13 (15)
Vomiting (Gastrointestinal disorders) | 4 (4) | 5 (6)
Fatigue (General disorders) | 5 (6) | 4 (4)
Nasopharyngitis (Infections and infestations) | 5 (5) | 3 (3)
Sinusitis (Infections and infestations) | 4 (4) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Balance disorder (Nervous system disorders) | 0 (0) | 4 (4)
Dizziness (Nervous system disorders) | 8 (9) | 18 (21)
Headache (Nervous system disorders) | 18 (20) | 16 (16)
Somnolence (Nervous system disorders) | 3 (3) | 5 (5)
Anxiety (Psychiatric disorders) | 4 (4) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.